CLINICAL TRIAL: NCT03731559
Title: Efficacy, Safety and Pharmacokinetics of Dolutegravir 50 Mg Once Daily with Food Versus Dolutegravir 50 Mg Twice Daily in HIV/TB Co-infected Patients Receiving Rifampin-based Antituberculosis Therapy
Brief Title: Efficacy, Safety and Pharmacokinetics of DTG with RIF
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Chest Division, Chulalongkorn University (Unknown); Infectious Disease, Chulalongkorn University (Unknown); Bamrasnaradura Infectious Diseases Institute (Other Government); Bhumibol Adulyadej Hospital (Other); Infectious Disease Taksin Hospital (Unknown); Klang Hospital (Unknown); Infectious Disease Chiangrai Prachanukroh Hospital (Unknown); Infectious Disease Chonburi Hospital (Unknown); Infectious Disease Buddhachinaraj Phitsanulok Hospital (Unknown); Radboud University Medical Center (Other); Ministry of Health, Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIV-NAT 254
Record Dates: First submitted 2018-10-31; First posted 2018-11-06 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: HIV/TB Coinfection
Keywords: Efficacy; safety; pharmacokinetics; Dolutegravir; HIV/TB co-infected patients; rifampin-based antituberculosis therapy
MeSH Terms: interventions — dolutegravir; Food; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DTG 50 mg OD with food (Active Comparator): DTG 50 mg OD with food plus 2NRTIs in HIV/TB co-infected patients receiving RIF based anti-TB therapy.
  Interventions: Drug: DTG 50 mg OD with food
- DTG 50 mg BID (Active Comparator): DTG 50 mg BID plus 2NRTIs in HIV/TB co-infected patients receiving RIF based anti-TB therapy.
  Interventions: Drug: DTG 50 mg BID

INTERVENTIONS:
Drug: DTG 50 mg OD with food — Dolutegravir 50 mg once daily with food plus 2NRTIs in HIV/TB co-infected patients receiving RIF based anti-TB therapy
  Arms: DTG 50 mg OD with food
Drug: DTG 50 mg BID — Dolutegravir 50 mg BID plus 2NRTIs in HIV/TB co-infected patients receiving RIF based anti-TB therapy.
  Arms: DTG 50 mg BID

SUMMARY:
The overall aim of the project is to evaluate optimal DTG dose for the combined treatment of TB and HIV infections with RIF based anti-TB therapy. This Stage II trial will determine precisely the PK parameters of DTG in combination with RIF regimen in Thai HIV/TB co-infected patients. After the optimal dose of DTG has been found, it will be further tested in a larger Stage III trial to assess its safety, tolerability and efficacy when used with RIF based regimen.

DETAILED DESCRIPTION:
This is a Stage II, randomized, open-label study describing the efficacy and safety of DTG 50 mg OD with food and DTG 50 mg BID plus 2NRTIs in HIV/TB co-infected patients receiving RIF based anti-TB therapy. The study will be conducted in approximately 200 HIV-1 infected individuals who are ART-naïve and newly diagnosed with probable or confirmed pulmonary, pleural, or lymph node (LN) Mycobacterium TB (MTB) taking RIF-containing first-line TB treatment. Subjects should have confirmed RIF-sensitive MTB infection as determined by GeneXpert (or equivalent approved molecular test) or mycobacterial culture.

The study is comprised two different stages:

1. Stage1, investigators will test the safety and tolerability, as well as Pharmacokinetics (PK), of two different doses of dolutegravir co-administered with standard anti-TB treatment. Overall, 40 HIV/TB patients will be enrolled. They will be randomized to 2 groups (DTG 50 mg with food and DTG 50 mg BID). Intensive PK of DTG will be performed at week 4. Interim analysis will be performed if all 40 cases completed 12 weeks and 24 weeks. Premature study termination will be set for

   1. proportion of HIV RNA < 50 copies/ml at week 24 between 2 group is different > 20%
   2. DTG 50 mg with food has geometric mean DTG Ctrough < 0.3 mg/L If there is no premature study termination met, the study will move to stage 2. Stage 2 will only be recruited if two different doses of dolutegravir are well tolerated and safe.
2. Stage 2: 160 HIV/TB patients will be enrolled. They will be randomized to 2 groups (DTG 50 mg with food and DTG 50 mg BID). DTG concentration will be performed at week 4 and 48. Interim analysis will be performed if all 200 cases completed 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. documented HIV positive
2. Aged >18 years
3. ARV naïve (previous exposure to ARV for < 2 weeks)
4. Any CD4 cell count
5. ALT <5 times ULN
6. estimated GFR>60 ml/min/1.73m2
7. Hemoglobin >7 mg/L
8. TB is diagnosed and there is a plan to receive stable doses of RIF containing anti-TB therapy for at least another 4 week period after initiation of ART
9. No other active OI (CDC class C event) except oral candidiasis or disseminated MAC
10. Body weight >40kg
11. Able to provide written informed consent

Exclusion Criteria:

1. Have documented history of HIV treatment failure or HIV mutation to NRTI, NNRTI, and/or INIs
2. Have previously treated for tuberculosis
3. Currently using immunosuppressive agents.
4. Currently using any prohibited medications that can affect the pharmacokinetics of the study drug such as phenobarbital, and carbamazepine
5. Currently using alcohol or illicit substances that may affect the conduct of the trial as per the opinion of the site Principal Investigator
6. Unlikely to be able to remain in the follow-up period as defined by the protocol
7. Patients with proven or suspected acute hepatitis. Patients with chronic viral hepatitis are eligible provided ALT, AST < 5 x ULN.
8. Have Karnofsky performance score <30%
9. Have TB meningitis, bone/joints (due to prolonged use of anti-TB drug)
10. Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-06-25 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
proportion of subjects from the ITT analysis population with plasma HIV-1 RNA <50 c/mL at Week 24 | Week 24
  The primary efficacy endpoint is the proportion of subjects from the ITT analysis population with plasma HIV-1 RNA <50 c/mL at Week 24.

SECONDARY OUTCOMES:
AUC of DTG concentration between DTG 50 mg with food OD and DTG 50 mg BID | Week 4
  AUC of DTG concentration between DTG 50 mg with food OD and DTG 50 mg BID
Cmax of DTG concentration between DTG 50 mg with food OD and DTG 50 mg BID | Week 4
  Cmax of DTG concentration between DTG 50 mg with food OD and DTG 50 mg BID
Cmin of DTG concentration between DTG 50 mg with food OD and DTG 50 mg BID | Week 4
  Cmin of DTG concentration between DTG 50 mg with food OD and DTG 50 mg BID
Oral clearance of DTG concentration between DTG 50 mg with food OD and DTG 50 mg BID | Week 4
  Oral clearance of DTG concentration between DTG 50 mg with food OD and DTG 50 mg BID
Proportion of subjects with plasma HIV-1 RNA <50 c/mL at Week 24 | Week 24
  Proportion of subjects with plasma HIV-1 RNA <50 c/mL at Week 24
Changes in CD4+ counts from baseline to Week 24 and Week 48 | Weeks 24 and 48
  Changes in CD4+ counts from baseline to Week 24 and Week 48
Incidence of disease progression | Week 48
  Incidence of disease progression (HIV-associated conditions, new AIDS diagnoses, and death)
Proportion of subjects that have completed TB treatment | Week 48
  Proportion of subjects that have completed TB treatment
Proportion of subjects that are cured from TB | Week 48
  Proportion of subjects that are cured from TB
Proportion of subjects that have relapsed | Week 48
  Proportion of subjects that have relapsed
Proportion of subjects that have defaulted | Week 48
  Proportion of subjects that have defaulted
TB outcome in terms of cure | Week 48
  Number of participants that have been cured of TB
TB outcome in terms of relapse | Week 48
  Number of participants with relapse
TB outcome in terms of treatment failure due to TB resistance | Week 48
  Number of participants with treatment failure due to TB resistance
TB outcome in terms of incidence | Week 48
  Incidence of all AEs, SAEs, and laboratory abnormalities
TB outcome in terms of severity | Week 48
  Severity of all AEs, SAEs, and laboratory abnormalities
discontinuation from the study | Week 48
  Proportion of subjects who permanently discontinued randomization arm due to AEs or death
discontinuation from the study drugs | Week 48
  Proportion of subjects who temporarily discontinued the study drugs and/or TB therapy due to AEs
Proportion of subjects with TB-associated IRIS | Week 48
  Proportion of subjects with TB-associated IRIS
AUC of DTG at Weeks 4 (with RIF) and 48 (without RIF) | Weeks 4 and 48
  AUC of DTG at Weeks 4 (with RIF) and 48 (without RIF) will be analyzed using population PK modeling approach to estimate AUC
Cmax of DTG at Weeks 4 (with RIF) and 48 (without RIF) | Weeks 4 and 48
  Cmax of DTG at Weeks 4 (with RIF) and 48 (without RIF) will be analyzed using population PK modeling approach to estimate Cmax
Ctrough of DTG at Weeks 4 (with RIF) and 48 (without RIF) | Weeks 4 and 48
  Ctrough of DTG at Weeks 4 (with RIF) and 48 (without RIF) will be analyzed using population PK modeling approach to estimate Ctrough
proportion of subjects with plasma HIV-1 RNA <50 c/mL at Week 48 | Week 48
  proportion of subjects with plasma HIV-1 RNA <50 c/mL at Week 48 (viral suppression)

CONTACTS AND LOCATIONS:
Overall Officials: Anchalee Avihingsanon, MD, PhD, Principal Investigator — HIV-NAT, Thai Red Cross - AIDS Research Centre
Locations (10):
- Thailand (10):
  - Klang Hospital, Bangkok, Bangkok
  - Bhumibol Adulyadej Hospital, Bangkok, Bangkok
  - Infectious Disease, Chulalongkorn University, Bangkok, Bangkok
  - Infectious Disease Taksin Hospital, Bangkok, Bangkok
  - Infectious Disease Chonburi Hospital, Chon Buri, Changwat Chon Buri
  - Bamrasnaradura Infectious Diseases Institute, Nonthaburi, Changwat Nonthaburi
  - Infectious Disease Buddhachinaraj Phitsanulok Hospital, Phitsanulok, Changwat Phitsanulok
  - Infectious Disease Chiangrai Prachanukroh Hospital, Chiang Rai, Chiangrai
  - Chest Division, Faculty of Medicine, Chulalongkorn University, Bangkok
  - HIV-NAT, Thai Red Cross - AIDS Research Centre, Bangkok